CLINICAL TRIAL: NCT02647411
Title: Increased Prevalence of Myopia in a Ophthalmologic Hospital in Goiânia - Goiás
Status: Completed | Type: Observational
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: ARVO R1 2016 1
Record Dates: First submitted 2015-11-11; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Myopia
Keywords: Prevalence; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Projeto Boa Visão: Review of records between 1995 and 2000, in totality of 16.806 patients between 2 and 40 years old
- Projeto Olhar Brasil: Review of records between March and September 2014, in totality of 163 patients between 6 and 18 years old

SUMMARY:
The purpose of this study was to evaluate the increased prevalence of myopia among patients in different periods in an ophthalmologic hospital in Goiania. There has been an increase of myopia prevalence around the world especially in some Asian countries. The investigators intend to analyze if this growing tendency is also present in our hospital, and if it exist how much is this growth.

DETAILED DESCRIPTION:
There were compared data collected in two scientific studies carried out in the same ophthalmologic hospital in different periods of time, they evaluated among other factors, the refractive errors of the participants, from this data there were compared the percentage of patients with myopia between the two studies. And analysed how much was the grown of myopia

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2 and 20 years assessment of Project "Olhar Brasil"
* Patients between 2 and 40 years assessment of Project "Boa visão"

Exclusion Criteria:

* The patients wasn't assessment of Project "Olhar Brasil"
* The patients wasn't assessment of Project "Boa Visão"

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 16.806 students from municipal schools of Goiânia during the period October 1995 to December 2000 In the second study there were selected 165 children from 2 to 14 years old who were referred to the Institute of Goiânia eyes, look at Brazil project within the school environment. The Look Brazil project aims to identify vision problems related to refraction.
Sampling Method: Non-Probability Sample
Enrollment: 16971 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Analisys of the percentage of patients with myopia in an ophthalmologic hospital in Goiânia - Goiás based on two prevalence studies made in the same hospital in different periods of time. | up to 2 months
  Comparison of the prevalence of myopia from data collected in two scientific studies carried out in the same ophthalmologic hospital in different periods of time, that evaluated among other factors the refractive errors of the participants.
  In the first study were examined 16.806 students from municipal schools of Goiania during the period October 1995 to December 2000. In the second study there were selected 165 children from 2 to 14 years old who were referred to the Institute of Goiânia eyes, by the "Projeto Boa Visão" within the school environment. The "Projeto Boa Visão" aims to identify vision problems related to refraction.